CLINICAL TRIAL: NCT06816225
Title: Association Between Sleep and Psychomotor Development in Early Childhood
Acronym: SleePsy
Status: Recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other); Up2Kids Pediatric Center - Vila Nova de Gaia (Unknown); USF Saúde no Futuro - Vila Nova de Gaia (Unknown)
Responsible Party: Sponsor
Other Study IDs: SleePsy
Record Dates: First submitted 2024-09-25; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-09

CONDITIONS: Sleep
Keywords: childhood,; psychomotor development; melatonin; actigraphy
MeSH Terms: interventions — Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy children: Aged 2 to 4 years old
  Interventions: Other: Actigraphy; Other: Schedule of Growing Skills II; Other: Questionnaire Children Sleep habits; Other: Melatonin evaluation

INTERVENTIONS:
Other: Actigraphy — Actigraphy is a validated complementary means of diagnosis, the gold standard for the assessment of circadian rhythm.
Other: Schedule of Growing Skills II — Assessment scale for skills in child development from 0 to 6 years.
Other: Questionnaire Children Sleep habits — Questionnaire for assessing sleep habits, validated for the Portuguese population (4) which allows us to understand the sleep hygiene habits of the child
Other: Melatonin evaluation — Melatonin will be measured in the first-morning urine and it is considered to be a good marker of plasma MLT level since its concentration is highly correlated with nocturnal plasma melatonin.

SUMMARY:
Sleep is a neurophysiological active process essential for healthy physical and cognitive development. In Portugal, there is no recent and objective data on how children sleep.

Given the importance of sleep in child health and development as well as the health gains achieved by establishing healthy sleep patterns since childhood, it seems extremely relevant to assess the various sleep parameters of Portuguese children and correlate them with their psychomotor and anthropometric development indicators. The results of this research work may support the implementation of sleep health education measures among parents, educators and policy makers, thus contributing to support the implementation of practices that promote sleep quality, napping until later in life as well as to promote the health of future adults.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 and 6 months year until the first assessment;
* Gestational age at birth 37 weeks or more;
* Delivery without serious complications for the child;
* Absence of developmental pathologies or pathologies that interfere with psychic and motor development;

Exclusion Criteria:

* Non-preterm birth but with severe growth restriction;
* Diagnosis of psychomotor development pathology;
* Diagnosis of pathology that interferes with psychomotor development;
* Taking daily medication, except vitamin supplements.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be healthy children aged 2 to 4 years old. Considering that the most prevalent differences in Growing Skills II scale scores will be around 3 and 5 points for a healthy toddler population as ours and that we will need to divide the population into 3 groups of sleep patterns (seriously sleep-restricted, moderately sleep-restricted and normal sleepers),
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep patterns | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  Sleep patterns based on movement tracking by sleep actigraphy.
Psychomotor development | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  The psychomotor developmental coefficient obtained through the application of the evaluation tool Schedule of growing skills II (SGS II) development scale.
Sleep hygiene | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  Sleep hygiene data obtained through the application of the Children Sleep habits questionnaire validated for the Portuguese population.
Melatonin levels | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  Levels of 6-sulphatoxymelatonin-aMT6, melatonin metabolite, measured in urine.

SECONDARY OUTCOMES:
Body Mass Index [BMI] | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  Weight [kg, kilogram] and height [m, meter] at the date of the evaluation for BMI-for-age calculation
Number of infectious events | At 24 - 30 months of age, at 3 years of age and at 4 years of age
  Number of infectious events in the first year of life and previous year of the following assessments.

OTHER OUTCOMES:
Demographics and lifestyle habits of the parents and family | At 24 - 30 months of age
  Questionnaire about demographic parameters and lifestyle of the parents and family:
  Age group (less than 24 years; 24-29; 30-35; 35-40; more than 40); Household; Level of education; Profession; Shift work; Smoking habits; Diet (omnivore, vegetarian, ovolactovegetarian, vegan or other); Average bedtime; Average total sleeping time; Sleep schedules between weekdays and the weekend; Chronotype; History of sleep disturbances; Vitamin supplementation during pregnancy; History of postpartum depression.
Medical history and biometrics of the child | At 24 - 30 months of age
  Questionnaire about the medical history and biometrics of the child:
  Gestational age at birth; APGAR index; Weight [kg, kilogram], length [meter, m] and head circumference [centimeter, cm] at birth; Type of feeding (breast milk, adapted milk or mixed feeding); Daycare attendance.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Keating, PhD, Principal Investigator — faculty of medicine
Locations (1):
- Faculty of Medicine (FMUP), Porto, Portugal